CLINICAL TRIAL: NCT04837703
Title: Managed Access Program (MAP) to Provide Access to Eltrombopag, for Treatment of Patients With Medically Significant Thrombocytopenia
Brief Title: MAP to Provide Access to Eltrombopag, for Treatment of Patients With Medically Significant Thrombocytopenia
Status: Available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CETB115B2003I
Record Dates: First submitted 2021-04-07; First posted 2021-04-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Thrombocytopenia
Keywords: Eltrombopag; thrombocytopenia; Idiopathic thrombocytopenic purpura; ITP; Severe aplastic anemia; SAA; HCV; Hepatitis C virus
MeSH Terms: conditions — Thrombocytopenia; Purpura, Thrombocytopenic, Idiopathic; Anemia, Aplastic; Hepatitis C | interventions — eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag should be taken at least two hours before or four hours after any products such as antacids, dairy products, or mineral supplements containing polyvalent cation (e.g. aluminum, calcium, iron, magnesium, selenium and zinc). Eltrombopag may be taken with food containing little (< 50 mg) or preferably no calcium.

SUMMARY:
The purpose of this Cohort Treatment Plan is to allow access to eltrombopag for eligible patients diagnosed with medically significant thrombocytopenia. The patient's Treating Physician should follow the suggested treatment guidelines and comply with all local health authority regulations.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this Treatment Plan have to meet all of the following criteria:

- Written informed consent must be obtained prior to any screening procedures or treatment assignment. If consent cannot be expressed in writing, it must be formally documented and witnessed, ideally via an independent trusted witness. An acceptable alternative (e.g., an assent form, or consent from a parent or guardian) should be signed for legally incompetent patients (e.g., children).

- In addition to informed consent, patients eligible for inclusion in this Treatment Plan may not be enrolled into any other eltrombopag clinical trial and must meet all of the following criteria (only one of the diseases listed under criterion No 1 is enough):

1. The patient must have any of the following diseases:

   * A confirmed diagnosis of chronic idiopathic thrombocytopenic purpura (ITP) according to the American Society of Haematology/ICR International consensus report on the investigation and management of primary immune thrombocytopenia reported by Neunert (2011) and Provan (2009), and the patient must be refractory to OR has relapsed after at least one prior ITP treatment recommended by the ASH/BCSH guidelines (corticosteroids or intravenous immunoglobulin (IVIg) or anti-D). Alternatively, a patient who is medically not eligible to receive corticosteroids must have had at least one alternative ITP treatment as recommended by the guidelines. Previous therapies for ITP and dates of administration must be recorded on the application form.
   * Severe aplastic anemia (SAA) patients who does not have an access to a comparable or satisfactory alternative treatment (i.e., comparable or satisfactory treatment is not available or does not exist).
   * HCV patients requiring treatment with an interferon based therapy and who have no access to alternative treatments.
2. The patient must have adequate medical condition and adequate organ function (e.g. renal, hepatic, cardiac function, etc.), as assessed by the treating physician.
3. Patients in childbearing age must be practicing an acceptable method of contraception from two weeks prior to administration of eltrombopag, throughout administration of eltrombopag, and 1 month after the last dose of eltrombopag.
4. Women of childbearing potential must have a negative serum pregnancy test within 14 days of first dose of program treatment and agree to use effective contraception, during the program and for one week following the last dose of program treatment.
5. The patient is able to understand and comply with all the requirements and instructions for receiving MAP

Exclusion Criteria:

Patients eligible for this Treatment Plan must not meet any of the following criteria:

1. Presence of moderate to severe impaired renal function as indicated by any or all of the following criteria:

   * Creatinine clearance < 45 mL/min as calculated using Cockcroft-Gault formula
   * Serum creatinine > 1.5 mg/dL
2. Total bilirubin > 1.5 × upper limit of normal (ULN)
3. Aspartate transaminase (AST) > 3.0 × ULN
4. Alanine transaminase (ALT) > 3.0 × ULN
5. Patient with liver cirrhosis.
6. Infection not adequately controlled with appropriate therapy.
7. Patients who are human immune deficiency virus (HIV), hepatitis C virus or hepatitis B surface antigen (HBsAg) positive. HCV-RNA negative patients are allowed to be enrolled.
8. Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient's ability to consent, be compliant with study procedures, tolerate protocol therapy, or patients with less than 3 months of life expectancy.
9. History of hypersensitivity to eltrombopag or to any of the excipients in eltrombopag
10. Patients with any prior history of arterial or venous thrombosis (stroke, transient ischemic attack, myocardial infarction, deep vein thrombosis or pulmonary embolism), AND ≥ two of the following risk factors: hormone replacement therapy, systemic contraception (containing oestrogen), smoking, diabetes, hypercholesterolemia, medication for hypertension, cancer, hereditary thrombophilic disorders (e.g., Factor V Leiden, ATIII deficiency, etc), or any other family history of arterial or venous thrombosis.
11. Patients with concurrent malignant disease.
12. Patients with SLE, antiphospholipid antibody syndrome or chronic hepatitis B infection,
13. Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions that could interfere with subject's safety, obtaining informed consent or compliance with the treatment guidelines.
14. Administration of an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of program treatment.
15. History of non-compliance with medical regimens or patients who are considered potentially unreliable and/or not cooperative, unwilling or unable to comply with the treatment guidelines.
16. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, (or female partners of male patients) unless they are using highly effective methods of contraception while taking study treatment and for 3 months after stopping medication. Highly effective methods of contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). For female patients on the study, the vasectomized male partner should be the sole partner for that patient
    * Use of oral (estrogen and progesterone), injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example, hormone vaginal ring or transdermal hormone contraception..
    * In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.
    * Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks in advance. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
17. Sexually active males must be willing to use a condom during intercourse while taking study treatment and for 3 months after stopping study treatment. A condom is required for all sexually active male participants to prevent them from fathering a child AND to prevent delivery of study treatment via seminal fluid to their partner. In addition, male participants must not donate sperm for the time period specified above.

If local regulations deviate from the contraception methods listed above to prevent pregnancy, local regulations apply and will be described in the informed consent form (ICF).

No additional exclusions may be applied by the investigator, in order to ensure that the study population will be representative of all eligible patients.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult